CLINICAL TRIAL: NCT06598332
Title: Administration of 5-Azacytidine With Steroids for First Line Therapy of Gastrointestinal GVHD
Brief Title: 5-Azacytidine With Steroids for Gastrointestinal GVHD (5-AZA FOR GVHD)
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: There is no funding.
Sponsor: Baylor College of Medicine (Other)
Collaborators: The Methodist Hospital Research Institute (Other); Center for Cell and Gene Therapy, Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, LaQuisa Hill, Assistant Professor, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-55921 5-AZA for GVHD
Record Dates: First submitted 2024-09-13; First posted 2024-09-19 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-08

CONDITIONS: Graft-Versus-Host Disease(GVHD)
Keywords: Graft-Versus-Host-Disease; GVHD; 5-AZACYTIDINE
MeSH Terms: conditions — Graft vs Host Disease | interventions — Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (Experimental): Patients will receive one cycle of AZA through the vein or as a shot under the skin daily for 5 days. This will start at the same time or within 3 days of starting standard treatment for gut GVHD with steroids.
  Interventions: Drug: 5-Azacytidine

INTERVENTIONS:
Drug: 5-Azacytidine — Patients will be treated with 5 azacytidine at a dose of 32 mg/m2 SQ or IV. The investigators aim to start AZA on Day 1 of steroids but it can be started up to 72 hours after steroids are started . Patients will be premedicated with antiemetics.
  Patients must receive steroids at a minimum dose of prednisone 2 mg/kg/day PO (or methylprednisolone 1.6 mg/kg/day IV) divided into 1-2 daily doses as therapy for acute GVHD. For patients that weigh over 100 kg, maximal starting dose of prednisone will be 200 mg (or methylprednisolone-equivalent).
  Steroid Taper for responding patients (Prednisone/Methylprednisolone) Days 1-5 2 mg/kg/day (taper cannot start until 3 days after enrollment) Days 6-10 1.5 mg/kg/day Day 11-15 1.0 mg/kg/day Days 16-20 0.5 mg/kg/day Days 21-28* 0.25 mg/kg/day Days 29-56 Gradual further taper with a goal of reaching < 0.2 mg/kg/day of prednisone (or < 0.16 mg/kg/day of methylprednisolone) by Day 56.

SUMMARY:
This study aims to evaluate the safety and feasibility of administering AZA in conjunction with steroids as first line therapy for GI GVHD.

A risk for patients who have received a transplant from another donor is graft versus host disease (GVHD). This happens because of differences between the donated cells (graft) and the patient body's cells (host). The new cells from the donor might see the patients body's cells as different and attack them. GVHD can be very serious and cause death. The standard first treatment for GVHD is corticosteroids but not all patients respond and they then have to receive other treatments. In addition, when GHVD involves the gut it can damage stem cells and can cause long term gut problems such as abdominal pain bowel disturbance. In laboratory studies giving a medicine called 5 -azacytidine (AZA) has been able to protect the gut stem cells and help them recover. In this trial the investigators would like to see if AZA can do the same thing when given with steroids in patients with GVHD.

Right now, doctors and researchers don't know the best treatment for GVHD. Acute GVHD is usually treated using high-dose corticosteroids, but these don't always work well. Even if the GVHD gets better when it involves the gut there can be long term damage to gut stem cells. In the laboratory 5 azacytidine (AZA) has been able to protect gut stem cells and help them recover and the investigators would like to learn if this happens in people too.

AZA has been approved by the U.S. Food and Drug Administration (FDA) for the treatment of patients with leukemias. It has also been used post transplant to try and risk the chance of leukemia coming back and to try and treat GVHD but AZA has not been approved by the FDA for the treatment of acute GVHD.

DETAILED DESCRIPTION:
Patients enrolled in this study will receive one cycle of AZA through the vein or as a shot under the skin daily for 5 days. This will start at the same time or within 3 days of starting standard treatment for gut GVHD with steroids

Medical tests before treatment--

Before being treated, patient will receive a series of standard medical tests:

* History and Physical exam
* Blood tests to measure blood cells, kidney and liver function
* A biopsy of the gut to look for GVHD is possible
* Serum pregnancy test for female patients who are of child bearing potential
* GVHD prophylaxis (prevention) medication
* Corticosteroid treatment
* An optional stool research sample

Medical tests during and after treatment--

Patient will receive standard medical tests when getting the GVHD treatment and afterwards:

* History and Physical exams
* Monitoring for GVHD
* Blood tests to measure blood cells, kidney and liver function
* A follow-up biopsy of the gut to look for GVHD is possible
* GVHD prophylaxis (prevention) medication
* Corticosteroid treatment
* Blood tests to measure blood cells, kidney and liver function
* Measurements of the tumor by routine imaging studies 6 weeks after the infusion.

To learn more about the way that AZA may work on gut stem cells an extra amount of blood will be obtained on the day AZA starts, 1, 2, 4, and 8 weeks after the T-cell infusion(s) and then at 3, 6 and 12 months. The amount of blood taken will be based on patient weight with up to a maximum of 60 mL (12 teaspoons) of blood to be obtained at any one time. This volume is considered safe, but may be decreased if patient is anemic (have a low red blood cell count).

If the patient has a repeat gut biopsy to check on their GVHD, investigators will request a sample to be used for research purposes.

Patients will receive supportive care for any acute or chronic toxicities, including blood components or antibiotics, and other intervention as appropriate.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 12 years of age or older at time of enrollment.
2. Patients experiencing their initial presentation of stage 1 or greater acute LGI GVHD requiring systemic therapy after allogeneic transplant for any malignant or non-malignant indication using any graft/donor source or conditioning intensity.
3. Patients can be enrolled with only a clinically established diagnosis. Biopsy of involved organs with acute GVHD is encouraged but is not required and should not delay study entry.
4. Patients should not have received systemic immune suppressive therapy for treatment of active GVHD except for a maximum of 72 hours of steroid therapy prior to enrollment. Topical skin and GI corticosteroids (such as budesonide and oral beclomethasone diproprionate) are allowed.
5. Informed Consent explained to, understood by and signed by patient/guardian. Patient/guardian given copy of informed consent.

Exclusion Criteria:

1. Relapsed, progressing or persistent malignancy or evidence of minimal residual disease (MRD) requiring withdrawal of systemic immune suppression.
2. Patients with acute GVHD developing after administration of a donor lymphocyte infusion (DLI) for relapse / progression of disease. Patients with acute GVHD after planned donor lymphocyte infusion or planned T cell or NK cell add back are eligible.
3. Patients with uncontrolled infections will be excluded. Infections are considered controlled if appropriate therapy has been instituted and, at the time of enrollment, no signs of progression are present. Progression of infection is defined as hemodynamic instability attributable to sepsis, new symptoms, worsening physical signs or radiographic findings attributable to infection. Persisting fever without other signs or symptoms
4. Patients receiving other drugs for the treatment of GVHD. Note, GVHD prophylaxis agents (e.g., calcineurin inhibitors) may be continued at local Investigator's discretion.
5. Patients on renal replacement therapy.
6. Patients requiring continuous supplemental oxygen (O2 requirement >2L/min to maintain peripheral O2 saturation [SpO2] >90%).
7. Patients with active hepatic sinusoidal obstructive syndrome (SOS) and/or clinical evidence of impaired hepatic function (ascites or encephalopathy related to liver disease)
8. Abnormal coagulation parameters (PT > 15 seconds, PTT > 40 seconds, and/or INR >1.5)
9. Significant active cardiac disease within the previous 6 months including:

   NYHA class 4 CHF Unstable angina Myocardial infarction
10. Known or suspected hypersensitivity to azacytidine.
11. Platelets <20 and or absolute neutrophil count (ANC) < 1000.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-08 (Estimated); Primary Completion 2028-05-01 (Estimated); Study Completion 2029-05-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility rate | 30 days after first dose of AZA
  The proportion of patients who can tolerate and complete one cycle of AZA (5-day) in combination with steroid among patients who are eligible and receive at least one dose of AZA.
Treatment-related adverse event (tAE) rate | 30 days after first dose of AZA
  The proportion of patients who develop any Grade 3-5 adverse events (per Common Terminology Criteria for Adverse Events [CTCAE] Version 5.0) that are considered probably, or definitely related to AZA or AZA in combination with steroid that occur in the first cycle of combination therapy until 30 days after first dose of AZA.

SECONDARY OUTCOMES:
GVHD response rate | Day 28
  The proportion of patients who have complete and partial response in patients who received steroids in combination with azacytidine.
Overall survival (OS) | 6 months and 12 months after combination therapy initiation
  Overall survival (OS) will be evaluated at 6 months and 12 months after combination therapy initiation. An event for OS is death from any cause.
Progression-free survival (PFS) | 6 months and 12 months after combination therapy initiation
  Progression-free survival (PFS) will be evaluated at 6 months and 12 months after combination therapy initiation. An event for PFS is death from any cause or relapse/progression of the primary disease.
Systemic Infections | 30 days after last dose of AZA
  The incidence of Grade 2 to 3 systemic infections (per BMT CTN Infection MOP), until 30 days after last dose of AZA will be described.

CONTACTS AND LOCATIONS:
Overall Officials: Helen Heslop, MD, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Houston Methodist Hospital, Houston, Texas
  - Texas Children's Hospital, Houston, Texas